CLINICAL TRIAL: NCT02638402
Title: Expression of Altered Glycosyltransferases, Mucins, and RTKs in Human Ovarian and Endometrial Cancers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201405068RINA
Record Dates: First submitted 2015-12-20; First posted 2015-12-23 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Carcinogenesis; Ovarian Cancer; Endometrial Cancer
Keywords: glycosylation; mucin; receptor tyrosin kinases; ovarian cancer; endometrial cancer
MeSH Terms: conditions — Carcinogenesis; Ovarian Neoplasms; Endometrial Neoplasms; Medullary cystic kidney disease 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stage I, II, III, IV ovarian cancer: Stage I, II, III, IV ovarian cancer receive treatment in National Taiwan University Hospital
- Stage I, II, III, IV endometrial cancer: Stage I, II, III, IV endometrial cancer receive treatment in National Taiwan University Hospital

SUMMARY:
To clarify the critical role of glycosyltransferases, altered Mucins, and RTKs in human ovarian and endometrial neoplasms, the study will examine the immunohistochemical expression profiles of glycosyltransferases, Mucins and receptor tyrosin kinases (RTKs) family in various stages and/or histologic subtypes of human ovarian and endometrial neoplasms and tissue microarrays.

DETAILED DESCRIPTION:
Glycosylation is a widely utilized chemical modification of proteins and lipids in mammalian cells during which saccharide units are covalently attached to the target structures and then sequentially elongated and branched - reactions facilitated by a large number of various glycosyltransferases. Alterations in this process have been associated with malignant transformation. To clarify the critical role of glycosyltransferases, altered Mucins (MUC), and RTKs in human ovarian and endometrial neoplasms, the study will examine the immunohistochemical expression profiles of glycosyltransferases (including β-1,4-Galactosyltransferase 1 (B4GALT1), β-1,4-Galactosyltransferase 3 (B4GALT3), β-1,4-N-Acetyl-Galactosaminyl Transferase 3 (B4GALNT3), Polypeptide N-Acetylgalactosaminyltransferase 2 (GALNT2), Polypeptide N-Acetylgalactosaminyltransferase 6 (GALNT6), β1,4-N-acetylglucosaminyltransferase III (GlcNAcT-III), β1,4-N-acetylglucosaminyltransferase V (GlcNAcT-V), and Glycoprotein-N-Acetylgalactosamine 3-Beta-Galactosyltransferase 1 (C1GALT1), Mucins (including MUC1, MUC3, MUC15, and MUC20) and receptor tyrosin kinases (RTKs) family (including epidermal growth factor receptor (EGFR), Src, VEGFR, and c-Met) in various stages and/or histologic subtypes of human ovarian and endometrial neoplasms and tissue microarrays, and compare them with clinicopathologic factors including outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian and endometrial cancer patients receiving operation in National Taiwan University Hospital

Exclusion Criteria:

* Recurrence or non-operable patients

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian and endometrial cancer patients receiving operation in National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Measure the Immunohistochemistry (IHC) expression | 5 years after patient received surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hau Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No